CLINICAL TRIAL: NCT00099905
Title: A Clinical Study to Assess the Efficacy and Safety of Three Doses of Vildagliptin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2301
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of three doses of vildagliptin, an unapproved drug, compared to placebo in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) in the range 22-45
* Blood glucose criteria must be met
* Not currently on drug therapy for type 2 diabetes

Exclusion Criteria:

* Type 1 diabetes
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c <7% after 24 weeks
Patients with reduction in HbA1c>/=to 0.7% after 24 weeks
Change from baseline in body weight at 24 weeks
Change from baseline in fasting lipids at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Pratley RE, Schweizer A, Rosenstock J, Foley JE, Banerji MA, Pi-Sunyer FX, Mills D, Dejager S. Robust improvements in fasting and prandial measures of beta-cell function with vildagliptin in drug-naive patients: analysis of pooled vildagliptin monotherapy database. Diabetes Obes Metab. 2008 Sep;10(10):931-8. doi: 10.1111/j.1463-1326.2007.00835.x. Epub 2007 Dec 17. PMID 18093207
- [Derived] Pratley RE, Rosenstock J, Pi-Sunyer FX, Banerji MA, Schweizer A, Couturier A, Dejager S. Management of type 2 diabetes in treatment-naive elderly patients: benefits and risks of vildagliptin monotherapy. Diabetes Care. 2007 Dec;30(12):3017-22. doi: 10.2337/dc07-1188. Epub 2007 Sep 18. PMID 17878242